CLINICAL TRIAL: NCT05777278
Title: A Prospective Study of Savolitinib Plus Docetaxel in Pretreated EGFR/ALK/ROS1/MET ex14m-wildtype Advanced NSCLC Patients With MET Overexpression (FirstMET)
Brief Title: Savolitinib Plus Docetaxel as 2L in EGFR/ALK/ROS1/MET ex14m-wildtype NSCLC With MET Overexpression
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FirstMET (ESR-22-21748)
Record Dates: First submitted 2023-02-21; First posted 2023-03-21 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Savolitinib; Docetaxel; MET Overexpression; Advanced NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; Docetaxel

STUDY DESIGN:
Intervention Model Description: Clinical trials with a single arm
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Savolitinib Plus Docetaxel (Experimental): Single Arm
  Interventions: Drug: Savolitinib; Drug: Docetaxel

INTERVENTIONS:
Drug: Savolitinib — Savolitinib (300mg or 200mg according to safety run-in recommendation, p.o., BID)
Drug: Docetaxel — Docetaxel (60 mg/m2, ivgtt, q3w)

SUMMARY:
This is a prospective, pilot, single-arm, single-center study exploring the efficacy and safety of savolitinib plus docetaxel as second-line therapy in patients with MET overexpressed, EGFR/ALK/ROS1/MET ex14m-wildtype advanced NSCLC.

Participants will receive treatment of docetaxel (60 mg/m2, ivgtt, q3w) in combination with savolitinib (300mg or 200mg according to safety run-in recommendation, p.o., BID) after informed consent signed. Treatment will continue until either objective disease progression, unacceptable toxicity occurs, consent is withdrawn, other discontinuation criterion is met, or study completion.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Provision of signed and dated, written ICF prior to any mandatory study specific procedures, sampling, and analyses.
3. Female or males age ≥18 years at the time of signing the ICF.
4. Histologically or cytologically confirmed locally advanced or metastatic EGFR/ALK/ROS1/MET ex14m-wildtype NSCLC.
5. Has only received first line systemic treatment of non-targeted advanced NSCLC.

   * Prior MET inhibitor therapy is not allowed.
   * At least 28 days since last treatment.
6. MET overexpression as determined IHC on tumor tissue.

   * MET overexpression by IHC, 3+ in ≥50% of tumor cells
   * Local IHC results are acceptable.
7. WHO or Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 with no deterioration over the previous 2 weeks prior to baseline or day of first dosing and a minimum life expectancy of 12 weeks.
8. At least 1 lesion that can be accurately measured at baseline as ≥10 mm in the longest diameter (except lymph nodes, which must have short axis ≥15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and is suitable for accurate repeated measurements.
9. Adequate haematological function defined as:

   * Haemoglobin ≥9 g/dL (no transfusion in the past 2 weeks).
   * Absolute neutrophil count ≥1.5×10^9/L.
   * Platelet count ≥100,000/μL (no transfusion in the past 10 days)
10. Adequate liver function defined as:

    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 x the upper limit of normal (ULN) with total bilirubin (TBL) ≤ ULN
    * OR TBL >ULN to ≤1.5x ULN with ALT and AST ≤ ULN, alkaline phosphatase (ALP) ≤ 2.5x ULN
11. Adequate renal function defined as a serum creatinine <1.5 times the institutional ULN OR a glomerular filtration rate ≥50 mL/min, as assessed using the standard methodology at the investigating centre (eg, Cockcroft-Gault, Modification of Diet in Renal Disease or Chronic Kidney Disease Epidemiology Collaboration formulae, ethylenediaminetetraacetic acid clearance or 24-hour urine collection). Confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN.
12. Adequate coagulation parameters, defined as:

    -International Normalisation Ratio (INR) <1.5 and activated partial thromboplastin time <1.5 x ULN unless patients are receiving therapeutic anti coagulation which affects these parameters.
13. Patients with known tumor thrombus or deep vein thrombosis are eligible if clinically stable on low molecular weight heparin (LMWH) for ≥2 weeks.
14. Ability to swallow and retain oral medications.
15. Willingness and ability to comply with study and follow-up procedures.
16. Females of childbearing potential should be willing to use highly effective contraceptive measures, should not be breast feeding, and must have a negative pregnancy test if of childbearing potential or must have evidence of non-childbearing potential by fulfilling one of the following criteria at screening:

    Post-menopausal is defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments; women under the age of 50 years would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution; or women with documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy.
17. Male patients with a female partner of childbearing potential should be willing to use barrier contraception during the study and for 6 months following discontinuation of study drug. Patients should refrain from donating sperm from the start of dosing until 6 months after discontinuing study treatment.

Exclusion Criteria:

1. As judged by the investigator, active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of oral therapy (eg, ulcerative disease, uncontrolled nausea, vomiting, diarrhoea Grade ≥2, and malabsorption syndrome).
2. Any of the following cardiac diseases currently or within the last 6 months:

   * Unstable angina pectoris
   * Congestive heart failure (New York Heart Association [NYHA] ≥Grade 2)
   * Acute myocardial infarction
   * Stroke or transient ischemic attack
3. Uncontrolled hypertension (BP ≥150/95 mmHg despite medical therapy).
4. Mean resting correct QT interval (QTcF) >470 msec for women and >450 msec for men on screening obtained from 3 electrocardiograms (ECGs) or factors that may increase the risk of QTcF prolongation such as chronic hypokalaemia not correctable with supplements, congenital or familial long QT syndrome, or family history of unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval and cause Torsade de Pointes.
5. Any clinically important abnormalities in rhythm, conduction or morphology of resting electrocardiograms (ECGs), e.g. complete left bundle branch block, third degree heart block, second degree heart block, PR interval >250 msec.
6. Serious underlying medical condition at the time of treatment that would impair the ability of the patient to receive protocol treatment.
7. Wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) administered ≤28 days or limited field radiation for palliation ≤7 days prior to starting study drug or has not recovered from side effects of such therapy.
8. Major surgical procedures ≤28 days of beginning study drug or minor surgical procedures ≤7 days. No waiting is required following port-a-cath placement.
9. As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, including renal transplant, active bleeding diatheses or uncontrolled hypertension, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol.
10. Active hepatitis B (HBV) (positive HBV surface antigen [HBsAg] result) or hepatitis C (HCV). Patients with a past or resolved HBV or HCV infection are eligible if:

    * Negative for HBsAg and positive for hepatitis B core antibody [anti-HBc] or
    * Positive for HBsAg, but for >6 months have had normal transaminases and HBV DNA levels between 0 to 2000 IU/mL (inactive carrier state) and willing to start and maintain antiviral treatment for at least the duration of the study.
    * Patients with a past or resolved HBV infection must have monthly monitoring of ALT and HBV DNA
    * HBV DNA levels >2000 IU/mL but on prophylactic antiviral treatment for the past 3 months and will maintain the antiviral treatment during the study.
    * Patients with positive HCV antibody are eligible only if the polymerase chain reaction is negative for HCV ribonucleic acid.
11. Presence of other active cancers, or history of treatment for invasive cancer, within the last 5 years. Patients with Stage I cancer who have received definitive local treatment at least 3 years previously and are considered unlikely to recur are eligible. All patients with previously treated in situ carcinoma (ie, non-invasive) are eligible, as are patients with history of non-melanoma skin cancer.
12. Unresolved toxicities from any prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 at the time of starting study treatment/randomization with the exception of alopecia.
13. Spinal cord compression or brain metastases unless asymptomatic, stable, and not requiring steroids for at least 2 weeks prior to start of study intervention. Subjects with leptomeningeal metastases are ineligible.
14. Past medical history of ILD/pneumonitis, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
15. Known serious active infection including, but not limited to, tuberculosis, or human immunodeficiency virus (positive human immunodeficiency virus 1/2 antibodies).
16. History of liver cirrhosis of any origin and clinical stage; or history of other serious liver disease or chronic disease with relevant liver involvement, with or without normal LFTs, such as

    * Hemochromatosis
    * Alpha-1 Antitrypsin deficiency
    * Autoimmune hepatitis (AIH)
    * Primary sclerosing cholangitis (PSC)
    * Primary biliary cirrhosis (PBC)
    * Biopsy-confirmed Non-Alcoholic Steatohepatitis (NASH) with advanced fibrosis
    * Biopsy- confirmed Alcoholic Steatohepatitis with advanced fibrosis
    * Wilson's disease
    * Hepatocellular carcinoma
17. Known contraindications to docetaxel administration.
18. Known hypersensitivity to the active or inactive excipients of docetaxel or savolitinib or drugs with a similar chemical structure or class.
19. Women who are either pregnant or breast-feeding.
20. Patients with previous medical history of Stevens Johnson syndrome (SJS) and serious cutaneous toxicity.
21. Prior exposure to HGF/MET inhibitors, e.g., foretinib, crizotinib, cabozantinib, merestinib, onartuzumab, capmatinib, tepotinib, etc.
22. Patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be strong inducers of CYP3A4, strong inhibitors of CYP1A2, within 2 weeks of the first dose of study treatment will be excluded. Herbal preparations/medications are not allowed throughout the study. These herbal medications include, but are not limited to: St. John's wort, kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng. Patients should stop using these herbal medications 7 days prior to first dose of study drug (three weeks for St John's wort). All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects on CYP3A4 during the study and for 3 months later the last dose intake (detailed description in Appendix G).
23. Participation in another clinical study with a study interventional medication administered within five half-lives of the compound or 3 months, whichever is greater or investigational medicinal device administered in the last 30 days prior to randomisation/first dose of study intervention or concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
24. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
25. Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions and requirements.
26. For women only-Currently breastfeeding.
27. Previous enrolments in the present study.
28. Without civil capacity or with restricted civil capacity.
29. Any other reasons judged by the leading investigator to prevent the subject from participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
ORR (Objective Response Rate) | The analysis will occur at 12 weeks after last patient in.
  ORR (Objective Response Rate) is defined as the proportion of participants who confirmed CR (Complete Response) or PR (Partial response) as their best overall response based on Response Evaluation Criteria in Solid Tumors (RECIST)1.1 as assessed by the investigator.

SECONDARY OUTCOMES:
PFS (Progression-Free Survival) | The analysis will occur when 70% data maturity of PFS events (14 PFS events) is observed in each cohort, at approximately 9 months after last patient in.
  PFS (Progression-Free Survival) is defined as the time from the first dose of study intervention until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the patient withdraws from therapy or receives another anti-cancer therapy prior to progression.
DoR (Duration of Response) | The analysis will occur when 70% data maturity of PFS events (14 PFS events) is observed in each cohort, at approximately 9 months after last patient in.
  DoR (Duration of Response) is defined as the time from the date of first documented response until date of documented progression or death in the absence of disease progression (ie, date of PFS (Progression-Free Survival) event or censoring-date of first response+1).
DCR (Disease Control Rate) | The analysis will occur at 12 weeks after last patient in.
  DCR (Disease Control Rate) is defined as the number(percent)of subjects with at least one visit response of confirmed CR (Complete Response), PR (Partial Response) or SD (Stable Disease), based on Investigator assessment according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
OS (Overall Survival) | The analysis will occur when 70% data maturity of PFS events (14 PFS events) is observed in each cohort, at approximately 9 months after last subject in, up to a maximum of approximately 3 years after first subject in.
  OS (Overall Survival) is defined as the time from the start of treatment until death due to any cause. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxing He, M.D, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Department of Thoracic Surgery and Oncology, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China